CLINICAL TRIAL: NCT00943917
Title: Phase 2 Study of ITCA 650 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of ITCA 650 (Exenatide in DUROS) in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-02
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- ITCA 650 20 mcg/day (Experimental)
  Interventions: Other: ITCA 650
- ITCA 650 40 mcg/day (Experimental)
  Interventions: Other: ITCA 650
- Exenatide Injection (Active Comparator)
  Interventions: Drug: Exenatide Injection
- ITCA 650 20/20 (Experimental)
  Interventions: Other: ITCA 650
- ITCA 650 20/60 (Experimental)
  Interventions: Other: ITCA 650
- ITCA 650 40/40 (Experimental)
  Interventions: Other: ITCA 650
- ITCA 650 40/80 (Experimental)
  Interventions: Other: ITCA 650
- Ex Inj/ITCA 650 40 (Experimental)
  Interventions: Other: Ex Inj/ITCA 650
- Ex Inj/ITCA 650 60 (Experimental)
  Interventions: Other: Ex Inj/ITCA 650

INTERVENTIONS:
Other: ITCA 650 — ITCA 650 (continuous delivery of exenatide in DUROS)
  Arms: ITCA 650 20 mcg/day; ITCA 650 20/20; ITCA 650 20/60; ITCA 650 40 mcg/day; ITCA 650 40/40; ITCA 650 40/80
Drug: Exenatide Injection — twice daily (BID) injections of exenatide commercially available Byetta: 5 mcg/dose first 12 weeks then 10 mcg/dose for 8 weeks
  Other Names: Byetta
  Arms: Exenatide Injection
Other: Ex Inj/ITCA 650 — twice-daily (BID) exenatide injection: 5 mcg/dose for 4 weeks then 10 mcg/dose for 8 weeks, followed by ITCA 650
  Other Names: Byetta
  Arms: Ex Inj/ITCA 650 40; Ex Inj/ITCA 650 60

SUMMARY:
The purpose of this study is to determine safety, efficacy and tolerability of various doses of ITCA 650 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18-70 years
* Type 2 diabetes mellitus for ≥ 6 months prior to Screening Visit 1
* On a stable (> 3 months prior to Screening Visit 1) treatment regimen of metformin monotherapy;
* Fasting plasma glucose < 240 mg/dL at Screening Visit 1
* HbA1c ≥ 7% and ≤ 10% at Screening Visit 1

Exclusion Criteria:

* Prior treatment with exenatide
* Treatment with any of the following antidiabetic agents within 3 months prior to Screening Visit 1: TZDs, sulfonylureas, DPP IV inhibitors, acarbose, or insulin (injected or inhaled)
* History of type 1 diabetes and/or history of diabetic ketoacidosis
* Body mass index ≥ 40 kg/m2;
* History of organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Study Site, Chino, California
  - Study Site, La Jolla, California
  - Study Site, National City, California
  - Study Site, Sacramento, California
  - Study Site, San Diego, California
  - Study Site, Valley Village, California
  - Study Site, Longmont, Colorado
  - Study Site, Pueblo, Colorado
  - Study Site, Bradenton, Florida
  - Study Site, Miami, Florida
  - Study Site, Miramar, Florida
  - Study Site, Pembroke Pines, Florida
  - Study Site, St. Petersburg, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Sandy Springs, Georgia
  - Study Site, Meridian, Idaho
  - Study Site, Chicago, Illinois
  - Study Site, Avon, Indiana
  - Study Site, Wichita, Kansas
  - Study Site, Lexington, Kentucky
  - Study Site, New Orleans, Louisiana
  - Study Site, Kalamazoo, Michigan
  - Study Site, Traverse City, Michigan
  - Study Site, Troy, Michigan
  - Study Site, Ypsilanti, Michigan
  - Study Site, Minneapolis, Minnesota
  - Study Site, Las Vegas, Nevada
  - Study Site, New Hyde Park, New York
  - Study Site, Charlotte, North Carolina
  - Study Site, Hickory, North Carolina
  - Study Site, Cincinnati, Ohio
  - Study Site, Franklin, Ohio
  - Study Site, Kettering, Ohio
  - Study Site, Norman, Oklahoma
  - Study Site, Eugene, Oregon
  - Study Site, Rapid City, South Dakota
  - Study Site, Austin, Texas
  - Study Site, Dallas, Texas
  - Study Site, Irving, Texas
  - Study Site, San Antonio, Texas
  - Study Site, West Jordan, Utah
  - Study Site, Norfolk, Virginia
  - Study Site, Olympia, Washington
  - Study Site, Spokane, Washington

REFERENCES:
- [Derived] Henry RR, Rosenstock J, Logan DK, Alessi TR, Luskey K, Baron MA. Randomized trial of continuous subcutaneous delivery of exenatide by ITCA 650 versus twice-daily exenatide injections in metformin-treated type 2 diabetes. Diabetes Care. 2013 Sep;36(9):2559-65. doi: 10.2337/dc12-2410. Epub 2013 May 3. PMID 23645886

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Stage II subjects divided into 6 total arms: ITCA 650 20 mcg/day assigned to either ITCA 650 20 mcg/day or ITCA 650 40 mcg/day; ITCA 650 40 mcg/day assigned to ITCA 650 40 mcg/day or ITCA 650 80 mcg/day; Ex Inj assigned to either ITCA 650 40 mcg/day or ITCA 650 60 mcg/day
Groups:
- ITCA 650 20 mcg/Day- STAGE I: ITCA 650 20 mcg/day continuous exenatide
- ITCA 650 40 mcg/Day- STAGE I: ITCA 650 40 mcg/day continuous exenatide
- Exenatide Injection- STAGE I: exenatide injection twice a day: 5 mcg/dose first 4 weeks then 10 mcg/dose for next 8 weeks
- ITCA 650 20/20- STAGE II: ITCA 650 20 mcg/day first 12 weeks, then ITCA 650 20 mcg/day through Week 24
- ITCA 650 20/60- STAGE II: ITCA 650 20 mcg/day first 12 weeks then ITCA 650 60 mcg/day through Week 24
- ITCA 650 40/40 - STAGE II: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 40 mcg/day through Week 24
- ITCA 650 40/80 - STAGE II: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 80 mcg/day through Week 24
- Ex Inj/ITCA 650 40 mcg/Day- STAGE II: Exenatide injection twice/day for 12 weeks then ITCA 650 40 mcg/day through Week 24
- Ex Inj/ITCA 650 60 mcg/Day- STAGE II: Exenatide injection twice/day for 12 weeks then ITCA 650 60 mcg/day through Week 24
- ITCA 650 20/20 Continuation: ITCA 650 20 mcg/day first 12 weeks then ITCA 650 through Week 48
- ITCA 650 20/40 Continuation: ITCA 650 20 mcg/day first 12 weeks then ITCA 650 40 mcg/day through Week 48
- ITCA 650 40/40 Contination: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 40 mcg/day through Week 48
- ITCA 650 40/80 Continuation: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 80 mcg/day through Week 48
- Ex Inj/ITCA 650 40 Continuation: Exenatide injection twice/day first 12 weeks then ITCA 650 40 mcg/day through Week 48
- Ex Inj/ITCA 650 60 Continuation: Exenatide injection twice daily first 12 weeks then ITCA 650 60 mcg/day through Week 48
Period: Stage I
Arm/Group | ITCA 650 20 mcg/Day- STAGE I | ITCA 650 40 mcg/Day- STAGE I | Exenatide Injection- STAGE I | ITCA 650 20/20- STAGE II | ITCA 650 20/60- STAGE II | ITCA 650 40/40 - STAGE II | ITCA 650 40/80 - STAGE II | Ex Inj/ITCA 650 40 mcg/Day- STAGE II | Ex Inj/ITCA 650 60 mcg/Day- STAGE II | ITCA 650 20/20 Continuation | ITCA 650 20/40 Continuation | ITCA 650 40/40 Contination | ITCA 650 40/80 Continuation | Ex Inj/ITCA 650 40 Continuation | Ex Inj/ITCA 650 60 Continuation
Started | 51 | 51 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 47 | 48 | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — hyperglycemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — A1C elevation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage II
Arm/Group | ITCA 650 20 mcg/Day- STAGE I | ITCA 650 40 mcg/Day- STAGE I | Exenatide Injection- STAGE I | ITCA 650 20/20- STAGE II | ITCA 650 20/60- STAGE II | ITCA 650 40/40 - STAGE II | ITCA 650 40/80 - STAGE II | Ex Inj/ITCA 650 40 mcg/Day- STAGE II | Ex Inj/ITCA 650 60 mcg/Day- STAGE II | ITCA 650 20/20 Continuation | ITCA 650 20/40 Continuation | ITCA 650 40/40 Contination | ITCA 650 40/80 Continuation | Ex Inj/ITCA 650 40 Continuation | Ex Inj/ITCA 650 60 Continuation
Started | 0 | 0 | 0 | 20 | 21 | 23 | 23 | 23 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 20 | 21 | 20 | 20 | 23 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage II Continuation
Arm/Group | ITCA 650 20 mcg/Day- STAGE I | ITCA 650 40 mcg/Day- STAGE I | Exenatide Injection- STAGE I | ITCA 650 20/20- STAGE II | ITCA 650 20/60- STAGE II | ITCA 650 40/40 - STAGE II | ITCA 650 40/80 - STAGE II | Ex Inj/ITCA 650 40 mcg/Day- STAGE II | Ex Inj/ITCA 650 60 mcg/Day- STAGE II | ITCA 650 20/20 Continuation | ITCA 650 20/40 Continuation | ITCA 650 40/40 Contination | ITCA 650 40/80 Continuation | Ex Inj/ITCA 650 40 Continuation | Ex Inj/ITCA 650 60 Continuation
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15 | 13 | 16 | 15 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 15 | 11 | 13 | 12 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — A1C elevation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ITCA 650 20 mcg/Day- STAGE I | ITCA 650 40 mcg/Day- STAGE I | Exenatide Injection- STAGE I | ITCA 650 20/20- STAGE II | ITCA 650 20/60- STAGE II | ITCA 650 40/40 - STAGE II | ITCA 650 40/80 - STAGE II | Ex Inj/ITCA 650 40 mcg/Day- STAGE II | Ex Inj/ITCA 650 60 mcg/Day- STAGE II | ITCA 650 20/20 Continuation | ITCA 650 20/40 Continuation | ITCA 650 40/40 Contination | ITCA 650 40/80 Continuation | Ex Inj/ITCA 650 40 Continuation | Ex Inj/ITCA 650 60 Continuation | Total
Number analyzed (Participants) | 51 | 51 | 53 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.3) | 53.3 (8.9) | 53.8 (9.6) |  |  |  |  |  |  |  |  |  |  |  |  | 53.7 (8.9)
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  |  |  | 0
  Between 18 and 60 years | 41 | 37 | 39 |  |  |  |  |  |  |  |  |  |  |  |  | 117
  >=60 years | 10 | 14 | 14 |  |  |  |  |  |  |  |  |  |  |  |  | 38
Gender [Number; unit: participants]
  Female | 26 | 28 | 24 |  |  |  |  |  |  |  |  |  |  |  |  | 78
  Male | 25 | 23 | 29 |  |  |  |  |  |  |  |  |  |  |  |  | 77
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 53 |  |  |  |  |  |  |  |  |  |  |  |  | 155

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1c (Per Protocol)
Description: Mean change in HbA1c over first 12 weeks (Stage I)
Time Frame: Day 0 and Week 12
Population: Per protocol analysis- Only subjects with values at baseline and Week 12 endpoint are included.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- ITCA 650 20 mcg/Day - STAGE I: ITCA 650 20 mcg/day through Week 12
- ITCA 650 40 mcg/Day - STAGE I: ITCA 650 40 mcg/day through Week 12
- Exenatide Injection - STAGE I: Exenatide injection twice daily: 5 mcg/dose first 4 weeks then 10 mcg/dose through Week 12
Arm/Group | ITCA 650 20 mcg/Day - STAGE I | ITCA 650 40 mcg/Day - STAGE I | Exenatide Injection - STAGE I
Number analyzed (Participants) | 47 | 45 | 47
percent change | -0.96 (0.905) | -1.04 (0.713) | -0.82 (0.870)

2. Primary Outcome: Mean Change in HbA1c (ITT)
Description: Mean change in HbA1c through Week 12
Time Frame: Day 0 to Week 12
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ITCA 650 20 mcg/Day - STAGE I | ITCA 650 40 mcg/Day - STAGE I | Exenatide Injection - STAGE I
Number analyzed (Participants) | 51 | 51 | 52
percent change | -.93 (0.882) | -0.96 (0.724) | -0.75 (0.866)

3. Primary Outcome: Mean Change in HbA1c (Per Protocol)
Description: Mean change in HbA1c through Week 24
Time Frame: Day 0 to Week 24
Population: Per protocol analysis - Only subjects with values at baseline and Week 24 endpoint are included.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- ITCA 650 20/20; ITCA 650 20/60; ITCA 650 40/40; ITCA 650 40/80; Ex Inj/ITCA 650 40; Ex Inj/ITCA 650 60: Stage II & Stage II Continuation
Arm/Group | ITCA 650 20/20 | ITCA 650 20/60 | ITCA 650 40/40 | ITCA 650 40/80 | Ex Inj/ITCA 650 40 | Ex Inj/ITCA 650 60
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 22 | 20
percent change | -.89 (.660) | -1.26 (.950) | -0.67 (.908) | -1.36 (0.664) | -1.01 (0.823) | -1.51 (1.266)

4. Primary Outcome: Mean Change in HbA1c (ITT)
Description: Mean change in HbA1c through Week 24
Time Frame: Day 0 to Week 24
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- ITCA 650 20/20: ITCA 650 20 mcg/day first 12 weeks then ITCA 650 20 mcg/day
- ITCA 650 20/60: ITCA 650 20 mcg/day first 12 weeks then ITCA 650 60 mcg/day
- ITCA 650 40/40: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 40 mcg/day
- ITCA 650 40/80: ITCA 650 40 mcg/day first 12 weeks then ITCA 650 80 mcg/day
- Ex Inj/ITCA 650 40: Exenatide injection first 12 weeks then ITCA 650 40 mcg/day
- Ex Inj/ITCA 650 60: Exenatide injection first 12 weeks then ITCA 650 60 mcg/day
Arm/Group | ITCA 650 20/20 | ITCA 650 20/60 | ITCA 650 40/40 | ITCA 650 40/80 | Ex Inj/ITCA 650 40 | Ex Inj/ITCA 650 60
Number analyzed (Participants) | 22 | 21 | 23 | 23 | 22 | 22
percent change | -0.89 (0.660) | -1.26 (0.950) | -0.70 (0.892) | -1.36 (0.664) | -1.01 (0.823) | -1.51 (1.266)

5. Primary Outcome: Mean Change in HbA1c (Per Protocol)
Description: Mean change in HbA1c through Week 48
Time Frame: Day 0 to Week 48
Population: Per protocol - Only subjects with values at baseline and Week 48 endpoint are included.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- ITCA 650 20/20: Stage II Continuation
Arm/Group | ITCA 650 20/20 | ITCA 650 20/60 | ITCA 650 40/40 | ITCA 650 40/80 | Ex Inj/ITCA 650 40 | Ex Inj/ITCA 650 60
Number analyzed (Participants) | 13 | 14 | 11 | 13 | 11 | 8
percent change | -1.00 (0.493) | -1.23 (0.908) | -0.69 (1.182) | -1.37 (0.837) | -1.45 (0.895) | -1.88 (1.212)

6. Primary Outcome: Mean Change in HbA1c (ITT)
Description: Mean change in HbA1c through Week 48
Time Frame: Day 0 to Week 48
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ITCA 650 20/20 | ITCA 650 20/60 | ITCA 650 40/40 | ITCA 650 40/80 | Ex Inj/ITCA 650 40 | Ex Inj/ITCA 650 60
Number analyzed (Participants) | 15 | 15 | 13 | 16 | 15 | 12
percent change | -1.13 (0.651) | -1.25 (0.880) | -0.48 (1.555) | -1.40 (0.803) | -1.16 (0.988) | -1.84 (1.570)

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- ITCA 650 20 mcg/Day: ITCA 650 20 mcg/day continuous exenatide
- ITCA 650 40 mcg/Day: ITCA 650 40 mcg/day continuous exenatide
- Exenatide Injection: exenatide injection twice daily dosing: 5 mcg/dose first 4 weeks then 10 mcg/day next 8 weeks
- ITCA 650 20/20 Continuation: ITCA 650 20 mcg/day first 12 weeks, then ITCA 650 20 mcg/day through Week 48
- ITCA 650 20/60 Continuation: ITCA 650 20 mcg/day first 12 weeks, then ITCA 650 60 mcg/day through Week 48
- ITCA 650 40/40 Continuation: ITCA 650 40 mcg/day first 12 weeks, then ITCA 650 40 mcg/day through Week 48
- ITCA 650 40/80 Continuation: ITCA 650 40 mcg/day first 12 weeks, then ITCA 650 80 mcg/day through Week 48
- Ex Inj/ITCA 40 Continuation: Exenatide twice/day first 12 weeks, then ITCA 650 40 mcg/day through Week 48
- Ex Inj/ITCA 650 60 Continutation: Exenatide injection first 12 weeks, then ITCA 650 60 mcg/day through Week 48
Arm/Group | ITCA 650 20 mcg/Day | ITCA 650 40 mcg/Day | Exenatide Injection | ITCA 650 20/20 | ITCA 650 20/60 | ITCA 650 40/40 | ITCA 650 40/80 | Ex Inj/ITCA 650 40 | Ex Inj/ITCA 650 60 | ITCA 650 20/20 Continuation | ITCA 650 20/60 Continuation | ITCA 650 40/40 Continuation | ITCA 650 40/80 Continuation | Ex Inj/ITCA 40 Continuation | Ex Inj/ITCA 650 60 Continutation
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/51 | 0/53 | 1/20 | 1/21 | 2/23 | 2/23 | 0/23 | 0/21 | 0/15 | 1/15 | 1/13 | 2/16 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 39/51 | 43/51 | 38/53 | 11/20 | 15/21 | 18/23 | 18/23 | 18/23 | 18/21 | 2/15 | 3/15 | 3/13 | 6/16 | 4/15 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ITCA 650 20 mcg/Day (N=51) | ITCA 650 40 mcg/Day (N=51) | Exenatide Injection (N=53) | ITCA 650 20/20 (N=20) | ITCA 650 20/60 (N=21) | ITCA 650 40/40 (N=23) | ITCA 650 40/80 (N=23) | Ex Inj/ITCA 650 40 (N=23) | Ex Inj/ITCA 650 60 (N=21) | ITCA 650 20/20 Continuation (N=15) | ITCA 650 20/60 Continuation (N=15) | ITCA 650 40/40 Continuation (N=13) | ITCA 650 40/80 Continuation (N=16) | Ex Inj/ITCA 40 Continuation (N=15) | Ex Inj/ITCA 650 60 Continutation (N=12)
cholecyctitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/19 (0) | 0/19 (0) | 0/22 (0) | 0/20 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/19 (0) | 1/19 (1) | 0/22 (0) | 0/20 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
meningitis cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/19 (0) | 1/19 (1) | 0/22 (0) | 0/20 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abortion, spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/19 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
subclavian artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/19 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITCA 650 20 mcg/Day (N=51) | ITCA 650 40 mcg/Day (N=51) | Exenatide Injection (N=53) | ITCA 650 20/20 (N=20) | ITCA 650 20/60 (N=21) | ITCA 650 40/40 (N=23) | ITCA 650 40/80 (N=23) | Ex Inj/ITCA 650 40 (N=23) | Ex Inj/ITCA 650 60 (N=21) | ITCA 650 20/20 Continuation (N=15) | ITCA 650 20/60 Continuation (N=15) | ITCA 650 40/40 Continuation (N=13) | ITCA 650 40/80 Continuation (N=16) | Ex Inj/ITCA 40 Continuation (N=15) | Ex Inj/ITCA 650 60 Continutation (N=12)
nausea (Gastrointestinal disorders) | 17 (19) | 24 (24) | 19 (20) | 2 (2) | 7 (8) | 1 (1) | 6 (7) | 1 (1) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 6 (6) | 9 (11) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 5 (7) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 4 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
early satiety (General disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
incision site hematoma (Injury, poisoning and procedural complications) | 8 (8) | 8 (8) | 0 (0) | 5 (5) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
incision site pruritis (Injury, poisoning and procedural complications) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
incision site hemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (6) | 3 (3) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
8 subjects (4 in 20, 1 in 40 and 3 in ex inj)completed StI but not randomized to St II; 3 subjects (2 in 20/20 & 1 in 40/80) who completed St I, randomized to St II but not given study drug. St II Cont was optional, so not all pts elected to continue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to submit multicenter results within 12 months after completion of the study. Thereafter, PI may publish the results of its data after submitting advance copy of the planned publication to sponsor. PI to agree to sponsor changes regarding deletion of confidential information, reasonable changes, or a delay of up to 90 days for patent purposes.